CLINICAL TRIAL: NCT05439850
Title: Arthroscopic Rotator Cuff Repair Augmented With Bioinductive Implant for Full-Thickness Tears: A Randomized Controlled Study
Brief Title: Bioinductive Patch for Full-Thickness Rotator Cuff Tears
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Stephanie Muh, MD, Deputy Service Chief, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15702
Record Dates: First submitted 2022-06-18; First posted 2022-06-30 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Tear Arthropathy
Keywords: Rotator Cuff Tear; Bioinductive; Arthroscopic Rotator Cuff Repair; Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Rotator Cuff Injuries; Rotator Cuff Tear Arthropathy | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of two groups. In the "control group," patients will receive the current surgical treatment for rotator cuff tears: debridement and repair. Patients in the "experimental group" will receive a bio-inductive patch following the same surgical treatment. Both groups of patients will participate in postoperative ultrasound imaging studies.
Who Masked: Participant
Masking Description: The study participant will not have knowledge of which treatment group he/she is randomized into for the duration of the study. Because the care provider/investigator will be required to implant the bioinductive patch, the physician will know into which treatment group each patient falls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Surgical treatment alone, consisting of arthroscopic rotator cuff repair. Ultrasound postoperatively at 1 year.
  Interventions: Procedure: arthroscopic rotator cuff repair; Diagnostic Test: Ultrasound Imaging
- Study Group (Experimental): Identical surgical treatment as control group plus bio-inductive patch implant. Ultrasound postoperatively at 1 year.
  Interventions: Procedure: arthroscopic rotator cuff repair; Biological: Bioinductive implant; Diagnostic Test: Ultrasound Imaging

INTERVENTIONS:
Procedure: arthroscopic rotator cuff repair — This procedure is the standard of care for rotator cuff tears who fail conservative treatment options.
Biological: Bioinductive implant — A bioinductive implant that is designed to promote healing of the torn rotator cuff tendon after surgery.
  Other Names: Bioinductive patch
  Arms: Study Group
Diagnostic Test: Ultrasound Imaging — An ultrasound will be performed on each patient one year postoperatively.

SUMMARY:
The purpose of this randomized-controlled study is to compare outcomes of arthroscopic rotator cuff repair augmented with a Bioinductive Implant (study group) to standard arthroscopic rotator cuff repair (control group). The primary outcome of this study is rotator cuff repair integrity (absence of full- or partial-thickness defect) demonstrated on ultrasound at 1-year postoperatively. The investigators hypothesize that the study group will have higher rates of repair integrity demonstrated on ultrasound at 1-year postoperatively.

DETAILED DESCRIPTION:
A bioinductive patch is an implant that may foster tendon regrowth and healing following surgery. Patients will be randomized into one of two groups: control and investigational. All surgical patients will have failed non-surgical/conservative options for 6 weeks. Patients in the "control group" will receive the standard surgery (arthroscopic rotator cuff repair) . Patients in the "experimental group" will receive the same surgical treatment, with the addition of the bioinductive patch. This patch will be implanted during surgery. Then, using a combination of ultrasound studies and other measures, the investigators will assess how well the patch works compared to surgery alone.

ELIGIBILITY:
Inclusion Criteria:

* Indicated and scheduled for arthroscopic rotator cuff repair.
* Full-thickness medium (1-3 cm), large (3-5 cm), and massive (>5 cm) rotator cuff tears involving the supraspinatus and/or infraspinatus tendons demonstrated on magnetic resonance or ultrasound imaging.
* Chronic, degenerative rotator cuff tears.
* Ability to read and understand English.
* Age ≥18 years
* Patient failed ≥6 weeks of conservative treatment, which included structured, in-person physical therapy or documented home therapy

Exclusion Criteria:

* Patient scheduled for open or mini-open rotator cuff repair
* Prior surgery of affected shoulder (except diagnostic arthroscopy)
* Partial-thickness rotator cuff tears
* Small (<1 cm) rotator cuff tears
* Rotator cuff tears involving the subscapularis tendon
* Acute and traumatic rotator cuff tears
* Active infection
* Cancer
* Autoimmune and rheumatologic disorders, including rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Rotator cuff repair integrity | Preoperative to 1 year postoperative
  absence of full- or partial-thickness defect as demonstrated on ultrasound at 1-year postoperatively.

SECONDARY OUTCOMES:
PROMs scores for upper extremity function | Preoperative to 2 years postoperative
  Patient-Reported Outcome Measures (PROMs) scores for upper extremity function. A T-score is given with a standard deviation based on the patients answers to the computerized adaptive test. The metrics have been designed to conform to a 0 - 100-point scale, with a score of 50 representing the mean of the population at large, 0 representing the minimum, and 100 representing the maximum function.
PROMs scores for depression | Preoperative to 2 years postoperative
  Patient-Reported Outcome Measures (PROMs) scores for depression. A T-score is given with a standard deviation based on the patients answers to the computerized adaptive test. The metrics have been designed to conform to a 10 - 90-point scale, with a score of 50 representing the mean of the population at large, 10 representing the minimum, and 90 representing the maximum function. A higher T-score represents higher increased depression (worse).
PROMs scores for upper extremity pain interference | Preoperative to 2 years postoperative
  Patient-Reported Outcome Measures (PROMs) scores for upper extremity pain and how it interferes with the patients daily life. A T-score is given with a standard deviation based on the patients answers to the computerized adaptive test. The metrics have been designed to conform to a 10 - 90-point scale, with a score of 50 representing the mean of the population at large, 10 representing the minimum, and 90 representing the maximum function. A higher T-score represents higher pain interference (worse).
Shoulder Range of Motion | Preoperative to 2 years postoperative
  Standard range of motion values collected by the surgeon during preoperative and followup visits
Shoulder Strength | Preoperative to 2 years postoperative
  Standard shoulder strength values collected by the surgeon during preoperative and followup visits. Medical Research Council Manual Muscle Testing scale will be used to measure the patient's strength on a 0 to 5 scale with 0 being the minimum and 5 being the maximum. Higher scores are better/normal.
Complications | Intraoperative to 2 years postoperative
  Both intra- and postoperative complications will be collected.
Reoperation | 2 years postoperative
  Whether or not patients required another operation.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J Muh, MC, Principal Investigator — Henry Ford Health
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.